CLINICAL TRIAL: NCT07263464
Title: The Association Between Tumor Necrosis Factor Superfamily Member 4 Polymorphism and Crohn's Disease
Brief Title: The Association Between TNFSF4 Polymorphism and CD
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-01-227
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Inflammatory Bowel Disease (Crohn's Disease and Ulcerative Colitis); Polymorphism, Single Nucleotide; Ustekinumab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Extract whole genome DNA from peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CD patients: Some CD patients received sufficient UST (6 mg/kg) intravenous infusion at week 0, followed by one subcutaneous (SC) dose of 90 mg UST at 8 weeks. Maintenance therapy consisted of 90 mg subcutaneous UST every 8 or 12 weeks.
  Interventions: Biological: Ustekinumab - Standard Dosage
- normal controls: no biological agents treatment

INTERVENTIONS:
Biological: Ustekinumab - Standard Dosage — Some CD patients received sufficient UST (6 mg/kg) intravenous infusion at week 0, followed by one subcutaneous dose of 90 mg UST at week 8.Maintenance therapy consisted of 90 mg subcutaneous UST every 8 or 12 weeks.
  Groups: CD patients

SUMMARY:
The goal of this observational study is to investigate the associations between tumor necrosis factor superfamily member 4 (TNFSF4) gene polymorphisms and the risk of Crohn's disease (CD), and to elucidate the impact of TNFSF4 gene variations on the CD clinical phenotype and the efficacy of ustekinumab (UST). The main question it aims to answer is: Does TNFSF4 polymorphism affect susceptibility to CD and the efficacy of UST in CD patients? Participants will have their blood drawn upon enrollment

DETAILED DESCRIPTION:
From January 2018 to May 2025, a total of 296 CD patients and 532 gender- and age-matched normal controls were collected from the Department of Gastroenterology, the Second Affiliated Hospital of Wenzhou Medical University.The genotypes of TNFSF4 were determined by multiplex polymerase chain reaction-ligase detection reaction technique. Unconditional logistic regression was employed to analyze the distribution of TNFSF4 gene polymorphisms between CD group and normal control group, as well as their influences on the clinicopathological characteristics of CD patients. Unconditional logistic regression model was used to explore the effect of TNFSF4 gene variation on the clinical response of CD patients in the treatment of UST at week 8 and mucosal healing at week 34, respectively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed CD based on comprehensive clinical, colonoscopy, histopathological, laboratory, and radiographic examination results

Exclusion Criteria:

* rheumatoid arthritis, systemic lupus erythematosus, intestinal tuberculosis, ischemic enteritis, radiation enteritis, tumors, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There was no statistically significant difference in the gender ratio, average age, and proportion of smokers between CD group and normal control group. All study subjects are from the Zhejiang Han population who are not related by blood.
Sampling Method: Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
the genotypes of TNFSF4 | Baseline
  multiplex polymerase chain reaction-ligase detection reaction technique

SECONDARY OUTCOMES:
clinical response of ustekinumab treatment | week 8
  the changes of the Crohn's disease activity index (CDAI)
clinical response of ustekinumab treatment | week 34
  the changes of the Crohn's disease activity index (CDAI)

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No